CLINICAL TRIAL: NCT07205861
Title: Auto-immune Thrombotic Thrombocytopenic Purpura : Retrospective Epidemiological Study of Patients in the National Cohort of the French TMA Center, TWI-LIGHT
Brief Title: Retrospective Epidemiological Study of Patients in the National Cohort of the French TMA Center
Acronym: TWILIGHT
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP240960
Record Dates: First submitted 2025-09-25; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-08

CONDITIONS: Thrombotic Thrombocytopenic Purpura (TTP); Immune Thrombotic Thrombocytopenic Purpura; Thrombotic Microangiopathies; Microangiopathy, Thromboic; Cardiovascular Diseases; Autoimmune Diseases; Rare Diseases; Neurological Manifestations
Keywords: Thrombotic Thrombocytopenic Purpura; Immune Thrombotic Thrombocytopenic Purpura; Thrombotic Microangiopathies (MeSH: D057049); Microangiopathies, Thrombotic (MeSH: D057172); ADAMTS13 Protein (MeSH: C423082); Autoimmune Diseases (MeSH: D001327); Cardiovascular Diseases (MeSH: D002318); Epidemiologic Studies (MeSH: D004812); Retrospective Studies (MeSH: D012196); Observational Study (Publication Type); Risk Factors (MeSH: D012307); Treatment Outcome (MeSH: D016647); Rare Diseases (MeSH: D034381); Longitudinal Studies (MeSH: D008159); Patient Registry (MeSH: D010329); Survival (MeSH: D009505); Quality of Life (MeSH: D011788); Neurological Manifestations (MeSH: D009462)
MeSH Terms: conditions — Purpura, Thrombotic Thrombocytopenic; Thrombotic Microangiopathies; Cardiovascular Diseases; Autoimmune Diseases; Rare Diseases; Neurologic Manifestations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- iTTP patients: The study is structured around one main cohort of all patients with immune thrombotic thrombocytopenic purpura (iTTP).
  Subgroup analyses are planned for specific populations: pregnant and postpartum women, pediatric patients, and elderly patients.
  There are no separate intervention or control groups; the design is a single retrospective cohort with multiple subgroup analyses.

SUMMARY:
Immune thrombotic thrombocytopenic purpura (iTTP) is a rare, life-threatening disorder characterized by microangiopathic hemolytic anemia, severe thrombocytopenia, and ischemic organ damage due to microvascular thrombosis. It results from a severe deficiency in the von Willeband factor (vWF)-cleaving protease ADAMTS13, primarily caused by autoantibodies that inhibit its activity. This deficiency leads to accumulation of ultra-large vWF multimers, triggering pathological platelet aggregation and widespread microthrombi. iTTP typically presents with acute neurological symptoms (e.g., confusion, seizures, coma), cardiac events (e.g., myocardial infarction), and multiorgan dysfunction. Without prompt treatment-plasma exchange, immunosuppression, and the vWF inhibitor caplacizumab-mortality exceeds 90%. Survivors face long-term risks, including cardiovascular complications, cognitive impairment, and reduced life expectancy.

The TWI-LIGHT protocol is a national retrospective epidemiological study coordinated by the French Reference Center for Thrombotic Microangiopathies (CNR-MAT). It aims to analyze long-term outcome in >1,200 iTTP patients diagnosed between October 2000 and June 2024. The study leverages pseudonymized data from the CNR-MAT registry, collected via a secure REDCap database.

Key Objectives:

1. Primary: Assess the impact of cardiovascular risk factors (e.g., hypertension, diabetes) and ADAMTS13 activity on life expectancy in iTTP survivors.
2. Secondary:

   * Evaluate disease burden in underrepresented groups (pregnant/postpartum women, children, elderly patients).
   * Analyze the influence of new therapies (caplacizumab, rituximab, recombinant ADAMTS13) on care pathways.
   * Identify prognostic factors and treatment practices.
   * Characterize neurocognitive outcomes and quality of life post-iTTP.

Methodology:

* Design: Non-interventional, retrospective (MR-004 compliance), using data from standard care.
* Inclusion: Patients with confirmed iTTP (thrombocytopenia, hemolytic anemia, ADAMTS13 <10%), diagnosed within the study period, and ≥1 year of follow-up.
* Exclusion: Cancer-associated iTTP, severe sepsis, or patient opposition to data reuse.
* Data Collection: Clinical, biological, and therapeutic variables from hospital/consultation records, including cardiovascular events, ADAMTS13 activity, and neurocognitive assessments.
* Analysis: Kaplan-Meier survival curves and Cox regression models to identify risk factors for non-iTTP-related death.

Expected Outcomes:

* Prevalence of cardiovascular comorbidities and their correlation with ADAMTS13 activity.
* Insights into iTTP subtypes (e.g., gestational, pediatric) and therapeutic efficacy.
* Evidence-based strategies for personalized long-term management.

Ethical Framework:

* AP-HP-sponsored, with oversight from Sorbonne University's ethics committee.
* Patients informed of data reuse with opt-out rights; data archived for 15 years.

This landmark study will inform clinical guidelines, optimize survivor care, and address unmet needs in iTTP management through comprehensive, real-world data analysis.

DETAILED DESCRIPTION:
The TWI-LIGHT protocol is a retrospective, non-interventional epidemiological study coordinated by the French National Reference Center for Thrombotic Microangiopathies (CNR-MAT). It leverages the CNR-MAT registry to analyze long-term outcomes in over 1,200 patients diagnosed with autoimmune thrombotic thrombocytopenic purpura (iTTP) between October 1, 2000, and June 1, 2024.

Background and Rationale iTTP is a rare, life-threatening disorder caused by severe ADAMTS13 deficiency, leading to microvascular thrombosis, multiorgan damage, and high mortality without prompt treatment. Survivors face long-term risks, including cardiovascular complications, cognitive impairment, and reduced life expectancy. Despite therapeutic advances (e.g., caplacizumab, rituximab), data on late complications, risk factors, and disease burden in underrepresented subgroups (e.g., pregnant women, children, elderly patients) remain limited. This study addresses critical gaps in understanding iTTP's natural history, treatment efficacy, and survival.

Study Design

* Type: Retrospective, multicenter, non-interventional (MR-004 compliance).
* Data Collected:

  * Acute Phase: Clinical presentation, lab results (standard biology, including ADAMTS13 activity, troponin), treatments (plasma exchange, immunosuppressants, caplacizumab).
  * Long-Term Follow-Up: Cardiovascular events (major adverse cardiovascular events, including ischemic stroke, myocardial infarction and angioplasty) and cardiovascular risk factors (hypertension, diabetes, weight and body mass index, dyslipidemia, smoking), ADAMTS13 activity trends, neurocognitive outcomes (quality-of-life scales: SF36, HADS), relapse rates, and mortality.
* Biobanking: ADAMTS13 samples stored at Hôpital Lariboisière (Prof. Veyradier's lab) under ethical approval (AC-2023-6021).

Expected Outcomes and Impact

* Clinical Insights:

  * Personalized cardiovascular risk profiles for iTTP survivors.
  * Evidence-based guidelines for pregnancy, elderly, and pediatric iTTP management.
  * Optimization of long-term monitoring (e.g., rituximab frequency).
* Health System Impact:

  * Cost-benefit analysis of novel therapies (e.g., caplacizumab, recombinant ADAMTS13).
  * Strategies to reduce diagnostic delays and hospitalizations. Real-World Relevance: Focus on underrepresented groups and long-term survival, with the goal to improve life expectancy of iTTP patients. This protocol represents a landmark effort to transform iTTP management through comprehensive real-world data, directly impacting clinical practice.
* Methodological Rigor: Centralized data auditing, ISO/IEC 17025-compliant biobanking.

ELIGIBILITY:
Inclusion Criteria:

-Patients with a diagnosis of immune mediated TTP

Exclusion Criteria:

* Cancer- associated iTTP and HIV-associated iTTP
* Severe sepsis
* Disseminated intravascular coagulation with consumption of coagulation factors;
* Transplant-associated TTP
* HIV-associated TTP (AIDS stage)
* Patient not affiliated with a social security scheme
* Patient or parent's objection to the reuse of their healthcare data for research

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of all patients in France diagnosed with thrombotic thrombocytopenic purpura (TTP), primarily the autoimmune subtype, between October 1, 2000, and June 1, 2024, who received care within the national network of the French Reference Center for Thrombotic Microangiopathies (CNR-MAT). This includes adults and children with autoimmune who have at least one year of follow-up. Patients are recruited from 6 core and 25 competence centers covering mainland France and overseas territories, ensuring nationwide representation. Data are collected from hospital and consultation records, and only patients who do not object to data reuse are included. This approach ensures a comprehensive, multicentric, and representative cohort for rare disease research.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2024-12-02 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
prevalence of major cardiovascular events | from diagnosis to last follow- up, up to 3 years
  ischemic strocke, myocardial infarction, reperfusion/angioplasty

SECONDARY OUTCOMES:
Incidence of cardiovascular risk factors | from diagnosis to last follow- up, up to 3 years
  Hypertension, diabetes, dyslipidaemia, smocking, body mass index,
correlation between ADMTS13 activity during remission and incidence of cardiovascular events and life expectancy | from remission to last follow- up, up to 3 years
characterization of pregnancy onset iTTP | from diagnosis to last follow- up, up to 3 years
  clinical presentation, management, prognosis(specific characteristics )
characterization of childhood onset iTTP | from diagnosis to last follow- up, up to 3 years
  clinical presentation, management, prognosis(specific characteristics )
characterization of elderly onset iTTP | from diagnosis to last follow- up, up to 3 years
  clinical presentation, management, prognosis(specific characteristics )

CONTACTS AND LOCATIONS:
Overall Officials: Paul COPPO, MD, PHD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Service d'Hématologie Hôpital Saint-Antoine, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided